CLINICAL TRIAL: NCT03946462
Title: A Prospective Randomized Controlled Trial of Supplemental Nitric Oxide During Cardiopulmonary Bypass to Reduce Acute Kidney Injury After Cardiac Surgery
Brief Title: Nitric Oxide During CPB to Reduce AKI in Neonates
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study could not be started because of some technical issues.
Sponsor: Fabio Savorgnan (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Fabio Savorgnan, Principal Investigator / Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-44435
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Congenital Heart Disease; Acute Kidney Injury
Keywords: Congenital Heart Disease; CHD; Acute Kidney Injury; AKI; Cardiopulmonary bypass; CPB; cardiac surgery; neonate; infant; nitric oxide; NO; gestational age
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: subjects, caregivers and research team members are blinded while respiratory therapists are unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NO Group (Experimental)
  Interventions: Drug: NO gas delivered during cardiac surgery
- Placebo Group (Placebo Comparator)
  Interventions: Other: placebo gas delivered during cardiac surgery

INTERVENTIONS:
Drug: NO gas delivered during cardiac surgery — intra-operative NO gas at 20ppm blended into the fresh gas flow of the CPB oxygenator via the INOMax delivery system.
  Arms: NO Group
Other: placebo gas delivered during cardiac surgery — placebo blended into the fresh gas flow of the CPB oxygenator via the INOMax delivery system. The placebo gas in this study will be 21% (or atmospheric) oxygen.
  Arms: Placebo Group

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled pilot study to investigate whether supplemental Nitric Oxide (NO) gas delivered during cardiac surgery with cardiopulmonary bypass (CPB) reduces the incidence and impact of acute kidney injury (AKI) in neonates undergoing surgery for congenital heart disease (CHD), when compared to placebo gas

DETAILED DESCRIPTION:
Screening: All patients undergoing either elective or emergency cardiac surgery will be screened against the eligibility criteria.

Research Sample Collection: Blood and urine will be collected for the first 48 hours admission and analyzed. The specific time points for these parameters will be: 2 hours, 6 hours, 12 hours 24 hours, and 48 hours post admission. Blood and urine parameters will also be collected as a baseline pre-operative. Patient outcomes will be captured for 30 days post operatively.

Research Data Collection: Baseline information will be collected. Other research related variables collected during the surgical intervention and bypass. Additional information will be collected 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours after admission as well as outcomes 30 days after the procedure.

Participants will be randomly allocated to the NO or control group in a 1:1 ratio.

This study is investigating a possible protective role for NO gas administration during bypass on the subsequent development of AKI. NO is typically delivered via large, stand-alone cylinders that are placed at the bedside (or adjacent to the patient) and is set up by respiratory therapists. In this research study, the study gas (NO or placebo) will be delivered directly into the bypass circuit at a constant gas flow. The placebo gas in this study will be 21% (or atmospheric) oxygen, and will appear to all members of the clinical and research teams (with the exception of the respiratory therapist responsible for setting it up) indistinguishable from NO, rendering this a double-blind study for the patient (or caregiver) and the investigators. This minimizes any possibility of bias in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: </= 30 days
* Gestational age: 38 weeks
* Diagnosis: Congenital Heart Disease (CHD)
* Planned surgery to include cardiopulmonary bypass (CPB )for underlying CHD
* Consent of parent/guardian

Exclusion Criteria:

* Currently receiving or has received inhaled nitric oxide (NO) or other nitrogen donors such as sildenafil or nitroprusside
* Pre-existing acute kidney injury (AKI) as per the AKIN criteria;
* Cardiac arrest within one week prior consent;
* Prior cardiac surgery with CPB procedure;
* Prior history of Extra Corporeal Membrane Oxygenation (ECMO)
* Use of another investigational drug.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
NGAL level | 48 hours
  1 of 2 biomarkers to determine acute kidney injury (AKI)
Cystatin-C level | 48 hours
  2 of 2 biomarkers to determine acute kidney injury (AKI)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Savorgnan, MD, Principal Investigator — Texas Children's Hospital / Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No